CLINICAL TRIAL: NCT02214446
Title: Explore Factors Related to Truth Telling in Primary Caregivers of Children Newly Diagnosed With Cancer
Brief Title: Factors Related to Truth Telling in Primary Caregivers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201311041RINC
Record Dates: First submitted 2013-12-10; First posted 2014-08-12 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Primary Caregivers of Children Newly Diagnosed With Cancer
Keywords: truth telling; hope; quality of life; care burden; children with cancer
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- primary caregivers of children newly diagnosed with cancer: Explore Factors related to Truth Telling in Primary Caregivers of Children Newly Diagnosed with Cancer

SUMMARY:
The purpose in this study was to investigate the current status, changes, correlation, and predictive factors of the truth telling, hope, care burden, and quality of life during treatment in primary caregivers of newly diagnosed children with cancer.

DETAILED DESCRIPTION:
Background: Over the last 50 years, telling truth in adult with cancer was direct. However, studies of truth telling in newly diagnosed children with cancer were seldom. Explore the factors and experiences related to truth telling in primary caregivers of children newly diagnosis with cancer were seldom too. Therefore, we could not estimate the current status of truth telling in primary caregivers of newly diagnosed children with cancer.

Purpose: The purpose in this study was to investigate the current status, changes, correlation, and predictive factors of the truth telling, hope, care burden, and quality of life during treatment in primary caregivers of newly diagnosed children with cancer.

Method: Purposive sampling structured questionnaire, used longitudinal resistance, repeated measurements, correlational design. SAS 9.3 for Windows was used for data entry and analyze. By using the frequency, percentage, mean, and standard deviation to describe demographic information and current status of truth telling. By using the mean, standard deviation, maximum and minimum to analyze hope, care burden, and quality of life. Demographic information, medical information data, truth telling, Herth Hope Index, caregiver burden scale, and quality of life index were tested by Pearson correlation coefficients; the change and predictors about truth telling, Herth Hope Index, caregiver burden scale, and quality of life index were tested by Generalized estimating equation.

Limitation: Studying in one medical center in Taipei, it could not estimate the country's primary caregivers of newly diagnosed children with cancer in conclusions. Because of the limitation of the manpower, time and case numbers, study tracked only six month, could not be assessed the long-term change of the Herth Hope Index, caregiver burden scale, truth telling and quality of life in primary caregivers of newly diagnosed children with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregivers of children newly diagnosed with cancer must be aged 20 years or older.
* Who can communicate in Chinese and Taiwanese.
* Consciousness clear.
* Normal cognitive function.
* After the explanation, agreed to participate in the study and signed a consent form.
* The age of children newly diagnosed with cancer is between 0 and 18 years old, who are newly diagnosed with cancer, before determined treatment plan.
* The physician of children newly diagnosed with cancer, who were willing to participate this study and signed a consent form.

Exclusion Criteria:

* Primary caregivers of children newly diagnosed with cancer, who have been diagnosed mental illness.
* The children were cancer recurrence.
* The physician of children newly diagnosed with cancer, who were not willing to participate this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Caregivers of Children Newly Diagnosed with Cancer
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
primary caregivers' Herth Hope Index | Change from baseline at family meeting at 3 months, and at 6 months
  The scores of primary caregivers' Herth Hope Index change from baseline at family meeting at 3 months, and at 6 months.
  We use Herth Hope Index(HHI) to evaluate the hope that the primary caregivers' care their child during treatment.
  There are twelve questions in the Herth Hope Index. The total score is from 12 to 48. Cronbach's α is .89. Retest is .80. Two weeks retest is .86.
  The higher the score is, the greater the hope is.
primary caregivers' quality of life index | Change from baseline at family meeting at 3 months, and at 6 months
  The scores of primary caregivers' quality of life index change from baseline at family meeting at 3 months, and at 6 months.
  We use quality of life index(Q.L.I) to evaluate the quality of life that the primary caregivers' care their child during treatment.
  There are 66 questions in the quality of life index. The total score is from 66 to 264. Cronbach's α is .95. Two weeks retest is .87.
primary caregivers' truth telling | Change from baseline at family meeting at 3 months, and at 6 months
  The primary caregivers' truth telling change from baseline at family meeting at 3 months, and at 6 months.
  Asking the primary caregivers' about that if you tell your child that he/she got the cancer, if you tell your child that he/she the treatment in future, and if you tell your child that he/she the rate of survival.
primary caregivers' care burden | Change from baseline at family meeting at 3 months, and at 6 months
  The scores of primary caregivers' care burden change from baseline at family meeting at 3 months, and at 6 months.
  We use Questionnaire of care burden to evaluate the care burde that the primary caregivers' care their child during treatment.
  There are 20 questions in the quality of life index. The total score is from 0 to 60. Cronbach's α is .91.
  The higher the score is, the heavier the care burden is.

CONTACTS AND LOCATIONS:
Overall Officials: SHIANN-TARNG JOU, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan